CLINICAL TRIAL: NCT06528067
Title: Mindful Motivation for Reducing Binge Eating
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Headspace Meditation Limited (Industry); National Center for Complementary and Integrative Health (NCCIH) (NIH); DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 23-40464; K23AT011048 (NIH)
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Binge Eating; Psychological; Health Behavior; Weight, Body
Keywords: Health; Meditation; Eating; Mindfulness; Students
MeSH Terms: conditions — Bulimia; Health Behavior; Body Weight | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Randomization in to one of two conditions:
  1. Mindful Motivation Intervention
  2. Active Control
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Motivation Group (Experimental): Participants will be assigned to a eating intervention that combines general mindfulness (via headspace) with motivational interviewing for mindful eating They will be asked to attend an online counseling session along with three 10-minute booster phone calls. They will be asked to engage with a digital-based mindful eating program once per week over the course of 8 weeks. In addition, participants will have access to optional educational materials on mindful eating and an optional online private support forum after the intervention period is finished.
  Interventions: Behavioral: Meditation; Behavioral: Mindful Motivation
- Active Control Condition (Active Comparator): Participants in the meditation intervention group will be assigned to a digitally-based meditation intervention (via Headspace) and asked to use this for at least 10 minutes a day over the course of 8 weeks.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — 10 minute per day, 8 week digital meditation
Behavioral: Mindful Motivation — A single 50 minute counseling session focused on eating behaviors, and three 10-minute follow-up phone calls to check-in on eating goals
  Arms: Mindful Motivation Group

SUMMARY:
The aim of this study is to test how acceptable and feasible a new eating intervention is in people with overweight and binge eating. This intervention combines mindful eating with motivational interviewing to target binge eating. The main questions this clinical trial aims to answer are:

How well do participants accept the new intervention (acceptability)? Is the intervention practical and easy to implement (feasibility)?

In this trial researchers will compare the new eating intervention (motivational interviewing for mindful eating + digital meditation) to an active control (digital meditation) to see if the intervention can help reduce binge eating.

Participants will:

1. Take online questionnaires at four different time points
2. Provide body composition and samples to measure glucose levels
3. Meditate for at least 10 minutes a day
4. If assigned to the Mindful Motivation group, 8 weeks of brief counseling

DETAILED DESCRIPTION:
In this clinical trial, researchers will recruit and randomize a total of 100 participants into an 8-week program. Participants will be assigned to either the 'Mindful Motivation' group (which combines motivational interviewing for mindful eating with digital meditation via headspace) or the 'Active Control' group (digital meditation via headspace only). Measurements will be taken at baseline, week 4, week 8 (post-intervention), and during a 6-month follow-up period. The researchers will look at changes in weight, waist circumference, glycated hemoglobin (A1C) levels, and continuous glucose levels for ten days (study 2 only, described below) at baseline and 8-week follow up.

Study 1: 40 participants will be adults from the community (20 in the intervention group and 20 in the active control group).

Study 2: 60 participants will be UCSF graduate students (30 in the intervention group and 30 in the active control group).

The Mindful Motivation program is adapted from several sources, including motivational interviewing for binge eating, motivational interviewing for weight management, and mindfulness-based eating awareness training (MB-EAT). The program includes an initial one-on-one counseling session, three booster calls during the 8-week intervention period, engagement with an online mindful eating program, instruction on mindful eating practices, access to an online anonymous support group, participation in an 8-week general mindfulness program (Headspace), and an optional 6-month follow-up with a counselor.

ELIGIBILITY:
Study 1

Inclusion Criteria:

* Aged 18 years or older
* Overweight (BMI ≥ 25 kg/m2)
* High levels of binge eating as assessed by QEWP-5 that are at least sub-clinical for binge eating disorder
* At least 1 episode of binge eating each month over the past 3 months with significant distress about these episodes
* Daily access to a smartphone or computer

Exclusion Criteria:

* Being an experienced meditator or having participated in a formal meditation practice in the last 3 months

Study 2

Inclusion Criteria:

* Current student at UCSF
* Aged 18 years or older
* Overweight (BMI ≥ 25 kg/m2)
* High levels of binge eating as assessed by QEWP-5 that are at least sub-clinical for binge eating disorder
* At least 1 episode of binge eating each month over the past 3 months with significant distress about these episodes
* Daily access to a smartphone or computer

Exclusion Criteria:

* Being an experienced meditator or having participated in a formal meditation practice in the last 3 months
* Inability to speak and read English or provide informed consent
* Significant medical or psychological concerns

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Client Satisfaction score, as determined by the total score on the Client Satisfaction Questionnaire (CSQ-8) | Mid-intervention to post-intervention, an anticipated average of 4 weeks
  The Client Satisfaction Questionnaire (CSQ-8) has a total score scale range of 8 to 32, with higher numbers indicating greater satisfaction
Change in Credibility/Expectancy and Satisfaction Questionnaire (CEQ) score, as determined by total score on the CEQ | Mid-intervention to post-intervention, an anticipated average of 4 weeks
  The CEQ consists of two subscales: credibility and expectancy. The CEQ contains 6 items rated on a 1-9 scale or a 0-100% scale depending upon the item. The first three and fifth items of the scale load onto the credibility factor and has a total score scale range of 4-36. The fourth and sixth item loads onto the expectancy factor and has a total score range of 2-22. The credibility score reflects how believable and convincing participants find the treatment, while the expectancy score reflects their expectations of how effective they think the treatment will be. Higher scores indicate greater credibility and higher expectations for the treatment's effectiveness.
Percentage of participants attending a phone call at the start of the intervention | Baseline
  By calculating the percentage of participants who attended the phone call at the start of the intervention the investigator aim to determine treatment feasibility. The higher the percentage of participants who attend the more feasible the intervention is for participants. The investigators aim for 80% attendance.
Percentage of participants attending a counseling session | Baseline
  By calculating the percentage of participants who attended the counseling session following the phone call the investigators aim to determine treatment feasibility. The higher the percentage of participants who attend the more feasible the intervention is for participants. The investigators aim for 80% attendance.
Percentage of participants attending a booster call # 1 | Mid intervention, an anticipated average of 1 week after counseling session
  By calculating the percentage of participants who attended the first booster call at mid intervention the investigators aim to determine treatment feasibility. The higher the percentage of participants who attend the more feasible the intervention is for participants. The investigators aim for 80% attendance.
Percentage of participants attending a booster call #2 | Mid intervention, an anticipated average of 2 week after first booster call
  By calculating the percentage of participants who attended the second booster call at mid intervention the investigator aim to determine treatment feasibility. The higher the percentage of participants who attend the more feasible the intervention is for participants. The investigators aim for 80% attendance.
Percentage of participants attending a booster call #3 | End if the intervention, an anticipated average of 3 weeks after the second booster call
  By calculating the percentage of participants who attended the third booster call at the end of the intervention the investigators aim to determine treatment feasibility. The higher the percentage of participants who attend the more feasible the intervention is for participants. The investigators aim for 80% attendance.

SECONDARY OUTCOMES:
Change in the Mindful Attention Awareness Scale (MAAS) questionnaire, as determined by the average score on the MAAS | Baseline to post-intervention, an anticipated average of 8 weeks
  The MAAS has a total average score scale range of 1 to 6, with higher numbers indicating greater dispositional mindfulness.
Change in self-reported motivation to change behavior, as determined by total score | Baseline to post-intervention, an anticipated average of 8 weeks
  This measure is composed of 3 questions, with each question ranging in score from 0 to 10, and total score scale range of 0 to 30, with higher numbers indicating motivation to change behavior. To see changes in motivation, 3 questions adapted from previous work (Miller and Rollnick, 2002) will be asked: "How important is it for the participant to change?" "How ready is the participant to change?" and If the participant decide to change, how confident is the participant that they will succeed?"
Change in Weight Efficacy Lifestyle Scale (WEL-SF) score, as determined by total score on the WEL-SF | Baseline to post-intervention, an anticipated average of 8 weeks
  The WEL-SF has a total score scale range of 1 to 88, with higher numbers indicating greater confidence in one's ability to resist overeating across 8 different scenarios.
Change in Reward Based Eating Drive Scale (RED-13) score, as determined by total score on the RED-13. | Baseline to post-intervention, an anticipated average of 8 weeks
  The RED-13 has a total score scale range of 13 to 65, with higher numbers indicating a greater drive to eat for reward or pleasure.
Change in Questionnaire on Eating and Weight Patterns (QEWP) frequency of binge eating episodes per month | baseline to post-intervention, an anticipated average of 8 weeks
  The first several items of the QEWP-5 assess the frequency of objectively large binge episodes (OBEs) per month. Frequency can range from 0 to 100+.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Radin, PhD, Principal Investigator — University of California, San Francisco; Elissa Epel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No